CLINICAL TRIAL: NCT04234776
Title: Intramuscular Ketamine Versus Escitalopram and Aripiprazole in Acute and Maintenance Treatment of Patients With Treatment-resistant Depression
Brief Title: Intramuscular Ketamine Versus Aripiprazole and Escitalopram in the Treatment of Resistant Depression
Acronym: KETProject
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Ricardo Alberto Moreno, M.D., Ph.D., Study principal investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: rampty2805
Record Dates: First submitted 2019-10-07; First posted 2020-01-21 (Actual); Last update posted 2020-01-21 (Actual); Status verified 2019-12

CONDITIONS: Depressive Disorder
Keywords: Ketamine; Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Treatment-Resistant | interventions — Ketamine; Escitalopram; Aripiprazole; Quality of Life

STUDY DESIGN:
Intervention Model Description: Subjects will receive IM ketamine or IM saline applications as randomized. Applications will occur three times a week. It will be 4 weeks of IM application (12 initial applications). Injections will occur into the subjects' glutes (0.75 mg / kg). The ketamine group will use 2 placebo tablets and the parallel group escitalopram 15 mg and aripiprazole 5 mg. Thereafter, participants will receive weekly ketamine doses over 6 months as maintenance treatment. Research members will be submitted to Structured Clinical Interview for the DSM for diagnostic categorization and will be evaluated from other scales. Vital signs will be checked continuously for a period of 2 hours with each infusion. Patients will be observed in a quiet, comfortable room and subjected to medical monitoring for 2 hours. They will leave the environment in the company of a competent adult.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rapid-acting antidepressant (Experimental): Subjects eligible to participate in the study will receive IM ketamine and will use 2 placebo tablets as randomized.
  Interventions: Drug: Ketamine; Diagnostic Test: Cognition; Other: Suicide risk; Other: Depression thoughts; Other: Quality of life and disability; Other: Clinical and epidemiological factors; Device: Safety of ketamine IM; Other: Tolerability of ketamine IM
- Comparator (Active Comparator): Subjects eligible to participate in the study will receive IM saline and will use escitalopram 15 mg and aripiprazole 5 mg as randomized
  Interventions: Drug: Ketamine; Diagnostic Test: Cognition; Other: Suicide risk; Other: Depression thoughts; Other: Quality of life and disability; Other: Clinical and epidemiological factors; Device: Safety of ketamine IM; Other: Tolerability of ketamine IM

INTERVENTIONS:
Drug: Ketamine — (0,75 mg/kg) saline solution (15 mg) Escitalopram (5 mg) Aripiprazole
  Other Names: Active comparator (escitalopram plus aripiprazole); Placebo
Diagnostic Test: Cognition — Composite tools
Other: Suicide risk — MADRS (10) and HAM-D (3)
Other: Depression thoughts — EPD
Other: Quality of life and disability — Quality of life and disability
Other: Clinical and epidemiological factors — Variables and categories
Device: Safety of ketamine IM — Vital signs
Other: Tolerability of ketamine IM — UKU-SERS, YOUNG, CADSS and BPRS-12.

SUMMARY:
The treatment of resistant depression should be optimized aiming at complete remission of symptoms, a complex condition due to several factors. Approximately 1/3 of patients with depressive disorders do not even respond to available antidepressants. Consequently, new molecules with robust action, fast effects and sustained improvement are currently being researched worldwide. Ketamine, an N-methyl-D-aspartate (NMDA) receptor antagonist, has emerged as a promising alternative due to its involvement in neurogenesis, synaptogenesis and consequent rapid improvement of depressive and suicidal symptoms with traditional intravenous (IV) use in sub dose (0.5 mg / kg). The therapeutic response of IV use has been short and requires monitoring in a hospital setting. There are no studies evaluating response to long-term ketamine use. Recent research has focused on identifying other routes of ketamine use such as intranasal and intramuscular (IM). The use of ketamine IM, despite the fact that there are few studies and small samples, can demonstrate efficacy in acute treatment and maintenance of depression, as well as low profile of side effects, greater accessibility potential, reduced costs and risks, patient comfort and possible expansion of resistant depression treatment capabilities in different settings.

DETAILED DESCRIPTION:
Compare the response of ketamine IM versus active control in treatment-resistant depression (TRD [primary outcome]) and find safety and tolerability of ketamine IM, evaluate changes in life quality, cognition and suicidal risk (secondary outcomes)

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of TRD, according to clinical evaluation and confirmed by SCID-IV (Structured Clinical Interview for the DSM);
2. Moderate to severe intensity of the disease;
3. Female patients in fertile conditions should be using a clinically accepted contraceptive method (oral contraceptive and/or condom);

   a. Blood test will be requested at the diagnostic stage and in case of clinical doubt as to the patient's gestational status,
4. Literate and able to understand the tasks requested;
5. With clinical comorbidities, however compensated;
6. Patients and/or legal representatives should understand the nature of the study and sign the Informed Consent Form.

Exclusion Criteria:

1. Imminent risk of suicide;
2. Patients with psychoactive substance dependence;
3. Intellectual deficit and psychotic symptoms;
4. Bipolar spectrum disorders and other primary psychiatric diagnoses;
5. Allergic to ketamine;
6. Glaucoma;
7. Treatment with reversible MAOI (monoamine oxidase inhibitor) in the week prior to visit 0;
8. Treatment with irreversible MAOI in two weeks prior to visit 0;
9. Fluoxetine treatment within 4 weeks prior to visit 0;
10. Treatment with others antidepressants;
11. Treatment with antipsychotics, lithium, benzodiazepines or other psychotropic drugs within 7 days prior to visit 0;

    a. Lorazepam and zolpidem may be used;
12. Patients who become pregnant will be excluded from the study and referred for obstetric care.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 88 (Estimated)
Dates: Start 2018-04-03 (Actual); Primary Completion 2020-06-03 (Estimated); Study Completion 2021-04-03 (Estimated)

PRIMARY OUTCOMES:
Change in depressive symptoms | 3 times a week in once month (Phase II)
  Montomery-Åsberg Depression Rating Scale ([0-60] higher scores: worse outcome). No improvement: MADRS ≤ 25% Partial response: MADRS ≥ 25% and < 50% Response: MADRS ≥ 50% Remission: MADRS ≤10
Change in depressive symptoms | Once a week in six months (Phase III)
  Montgomery-Åsberg Depression Rating Scale ([0-60] higher scores: worse outcome).
  Recovery: Maintenance ≥ 6-8 months Relapse: Full return of symptoms once remission has occurred or worsening ≤ 75% with lower percentage of improvement (HAM-D inclusion criteria)
Change in depressive symptoms | Once a week in once month (Phase IV)
  Montgomery-Åsberg Depression Rating Scale ([0-60] higher scores: worse outcome).
  Relapse: Full return of symptoms once remission has occurred or worsening ≤ 75% with lower percentage of improvement (HAM-D inclusion criteria).

SECONDARY OUTCOMES:
Depression symptoms | Through study completion, an average of 1 year.
  Hamiltom Depression Ratins Scale (HAM-D [0-50] higher scores: worse outcome).
Clinical impressions-S | Through study completion, an average of 1 year.
  Clinical Global Impression Scale (CGI [0-7] higher scores: worse outcome).
Clinical impressions-I | Through study completion, an average of 1 year.
  Clinical Global Impression Scale (CGI [0-7] higher scores: worse outcome).
Electrocardiographic monitoring | 3 times a week in once month (Fase II) and once a week in six months (Phase III)
  P wave, PR interval, QRS complex, J-point, ST segment, T wave, Corrected QT interval and U wave Rhythm (irregular rhythm: worse outcome).
Blood Pressure (BP [mmHg]). | 3 times a week in once month (Fase II) and once a week in six months (Phase III)
  BP low <90/60 (systolic/diastolic) mmHg and high >140/90 mmHg ( (systolic/diastolic).
Heart rate (HR [bpm]). | 3 times a week in once month (Fase II) and once a week in six months (Phase III)
  Anormal HR <60 bpm or >100 bpm.
Digital pulse oximetry (%). | 3 times a week in once month (Fase II) and once a week in six months (Phase III)
  Low oxygen saturation <95%.
Respiratory rate (RR [cycles/min]) | 3 times a week in once month (Fase II) and once a week in six months (Phase III)
  Anormal RR <10 cycles/min or >20 cycles/min.
Suicide risk 1 | Through study completion, an average of 1 year.
  Montgomery-Åsberg Depression Rating Scale (item 10 [0-6] higher scores: worse outcome).
Suicide risk 2 | Through study completion, an average of 1 year.
  Hamilton Depression Rating Scale (item 3 [0-4] higher scores: worse outcome).
General side effects | 3 times a week in once month (Phase II) and once a week in six months (Phase III)
  Ugvalg for Kliniske Undersgelser-Side Effect Rating Scale (UKU-SERS [48 specific symptoms).
Hypo/maniac symptoms | 3 times a week in once month (Phase II) and once a week in six months (Phase III)
  Young Mania Rating Scale (YOUNG [0-58] higher scores: worse outcome).
Dissociative symptoms | 3 times a week in once month (Phase II) and once a week in six months (Phase III)
  Clinician-Administered Dissociative State Scale (CADSS [0-108] higher scores: worse outcome)
Psychotic symptoms | 3 times a week in once month (Phase II) and once a week in six months (Phase III)
  Brief Psychiatric Rating Scale (item 12 [0-6] higher scores: worse outcome).
Depression thoughts | Through study completion, an average of 1 year.
  Depression Thoughts Scale (EPD [1-78] higher scores: worse outcome)
Stimate intelligence quocient | Through study completion, an average of 1 year.
  Wechsler Abreviated Scale of Intelligence (WASI [70-160 percentille] higher scores: better outcomes).
Intelligence quocient | Through study completion, an average of 1 year.
  Wechsler Scale of Intelligence (WAIS III [70-155 percentille] higher scores: better outcomes).
Attention | Through study completion, an average of 1 year.
  Trial Making Test (5-95 percentille, higher scores: better outcomes).
Memory | Through study completion, an average of 1 year.
  Rey figures (10-100 percentille, higher scores: better outcomes)
Executive functions 1 | Through study completion, an average of 1 year.
  Wisconsin Test (50->80 score, higher scores: better outcomes).
Executive functions 2 | Through study completion, an average of 1 year.
  Stroop Color Word Test (5-95 percentille, higher scores: better outcomes)
Verbal fluency 1 | Through study completion, an average of 1 year.
  Verbal Fluency Test (FAS [10-90 percentille], higher scores: better outcomes))
Verbal fluency 2 | Through study completion, an average of 1 year.
  The Rey Auditory-Verbal Learning Test (RAVLT [5-95 percentille], higher scores: better outcomes).
Functional recovery 1 | Through study completion, an average of 1 year.
  World Health Organization Quality of Life (WHOQOL-brief [4 domains, 26 questions higher scores: better outcome]).
Functional recovery 2 | Through study completion, an average of 1 year.
  Sheehan Disability Scale (SDS [0-30] higher scores: worse outcome).
Body Mass Index (BMI) | Through study completion, an average of 1 year.
  Weight and height (kg/m2).
Clinical and psychiatric features 1 | Through study completion, an average of 1 year.
  Disease intensity (HAM-D [% of patients], moderate or severe)
Clinical and psychiatric features 2 | Through study completion, an average of 1 year.
  Number of episodes (questionnaire [incidence])
Clinical and psychiatric features 3 | Through study completion, an average of 1 year.
  Current episode duration (questionnaire [years])
Clinical and psychiatric features 4 | Through study completion, an average of 1 year.
  Suicide attempts (questionnaire [% of pacients])
Clinical and psychiatric features 5 | Through study completion, an average of 1 year.
  History of physical abuse (questionnaire [% of pacients])
Clinical and psychiatric features 6 | Through study completion, an average of 1 year.
  History of sexual abuse (questionnaire [% of pacients])
Clinical and psychiatric features 7 | Through study completion, an average of 1 year.
  Psychiatric hospitalizations (questionnaire [% of pacients])
Clinical and psychiatric features 8 | Through study completion, an average of 1 year.
  Clinical comorbidities (questionnaire [% of patients]).
Clinical and psychiatric features 9 | Through study completion, an average of 1 year.
  Family history of depression (questionnaire [% of patients])
Clinical and psychiatric features 10 | Through study completion, an average of 1 year.
  Family history of bipolar disorders (questionnaire [% of patients)
Clinical and psychiatric features 11 | Through study completion, an average of 1 year.
  Family history of other mental disorders (questionnaire [% of patients]).
Epidemiological features 1 | Through study completion, an average of 1 year.
  Age (questionnaire [years]).
Epidemiological features 2 | Through study completion, an average of 1 year.
  Gender (questionnaire [% of patients]; male/female)
Epidemiological features 3 | Through study completion, an average of 1 year.
  Marital status (questionnaire [% of patients] single, married, separated, divorced or widower).
Epidemiological features 4 | Through study completion, an average of 1 year.
  Ethnicity (questionnaire [% of patients])
Epidemiological features 5 | Through study completion, an average of 1 year.
  Religion (questionnaire [% of patients] protestant, pentecostal or neopentecostal, spiritism, afro-brazilian, no religion or atheism and others]).
Epidemiological features 6 | Through study completion, an average of 1 year.
  Occupation (questionnaire [% of patients])
Epidemiological features 7 | Through study completion, an average of 1 year.
  Education (questionnaire [years])
Epidemiological features 8 | Through study completion, an average of 1 year.
  Individual income (questionnaire [dollars]).
Epidemiological features 9 | Through study completion, an average of 1 year.
  Family income (questionnaire [dollars]).

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A Moreno, MD, PhD, Principal Investigator — Department and Institute of Psychiatry, University of Sao Paulo
Locations (1):
- Núcleo de Pesquisas em Saúde Mental, Blumenau, Santa Catarina, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rush AJ, Trivedi MH, Wisniewski SR, Nierenberg AA, Stewart JW, Warden D, Niederehe G, Thase ME, Lavori PW, Lebowitz BD, McGrath PJ, Rosenbaum JF, Sackeim HA, Kupfer DJ, Luther J, Fava M. Acute and longer-term outcomes in depressed outpatients requiring one or several treatment steps: a STAR*D report. Am J Psychiatry. 2006 Nov;163(11):1905-17. doi: 10.1176/ajp.2006.163.11.1905. PMID 17074942
- [Result] Bennabi D, Aouizerate B, El-Hage W, Doumy O, Moliere F, Courtet P, Nieto I, Bellivier F, Bubrovsky M, Vaiva G, Holztmann J, Bougerol T, Richieri R, Lancon C, Camus V, Saba G, Haesbaert F, d'Amato T, Charpeaud T, Llorca PM, Leboyer M, Haffen E. Risk factors for treatment resistance in unipolar depression: a systematic review. J Affect Disord. 2015 Jan 15;171:137-41. doi: 10.1016/j.jad.2014.09.020. Epub 2014 Oct 8. PMID 25305428
- [Result] Philip NS, Carpenter LL, Tyrka AR, Price LH. Pharmacologic approaches to treatment resistant depression: a re-examination for the modern era. Expert Opin Pharmacother. 2010 Apr;11(5):709-22. doi: 10.1517/14656561003614781. PMID 20151847
- [Result] Kennedy SH, Lam RW, McIntyre RS, Tourjman SV, Bhat V, Blier P, Hasnain M, Jollant F, Levitt AJ, MacQueen GM, McInerney SJ, McIntosh D, Milev RV, Muller DJ, Parikh SV, Pearson NL, Ravindran AV, Uher R; CANMAT Depression Work Group. Canadian Network for Mood and Anxiety Treatments (CANMAT) 2016 Clinical Guidelines for the Management of Adults with Major Depressive Disorder: Section 3. Pharmacological Treatments. Can J Psychiatry. 2016 Sep;61(9):540-60. doi: 10.1177/0706743716659417. Epub 2016 Aug 2. PMID 27486148
- [Result] Saveanu R, Etkin A, Duchemin AM, Goldstein-Piekarski A, Gyurak A, Debattista C, Schatzberg AF, Sood S, Day CV, Palmer DM, Rekshan WR, Gordon E, Rush AJ, Williams LM. The international Study to Predict Optimized Treatment in Depression (iSPOT-D): outcomes from the acute phase of antidepressant treatment. J Psychiatr Res. 2015 Feb;61:1-12. doi: 10.1016/j.jpsychires.2014.12.018. Epub 2014 Dec 31. PMID 25586212
- [Result] Perlis RH. A clinical risk stratification tool for predicting treatment resistance in major depressive disorder. Biol Psychiatry. 2013 Jul 1;74(1):7-14. doi: 10.1016/j.biopsych.2012.12.007. Epub 2013 Feb 4. PMID 23380715
- [Result] McIntyre RS, Filteau MJ, Martin L, Patry S, Carvalho A, Cha DS, Barakat M, Miguelez M. Treatment-resistant depression: definitions, review of the evidence, and algorithmic approach. J Affect Disord. 2014 Mar;156:1-7. doi: 10.1016/j.jad.2013.10.043. Epub 2013 Nov 15. PMID 24314926
- [Result] Spielmans GI, Berman MI, Linardatos E, Rosenlicht NZ, Perry A, Tsai AC. Adjunctive atypical antipsychotic treatment for major depressive disorder: a meta-analysis of depression, quality of life, and safety outcomes. PLoS Med. 2013;10(3):e1001403. doi: 10.1371/journal.pmed.1001403. Epub 2013 Mar 12. PMID 23554581
- [Result] Millan MJ, Goodwin GM, Meyer-Lindenberg A, Ove Ogren S. Learning from the past and looking to the future: Emerging perspectives for improving the treatment of psychiatric disorders. Eur Neuropsychopharmacol. 2015 May;25(5):599-656. doi: 10.1016/j.euroneuro.2015.01.016. Epub 2015 Feb 7. PMID 25836356
- [Result] Ferrari AJ, Charlson FJ, Norman RE, Patten SB, Freedman G, Murray CJ, Vos T, Whiteford HA. Burden of depressive disorders by country, sex, age, and year: findings from the global burden of disease study 2010. PLoS Med. 2013 Nov;10(11):e1001547. doi: 10.1371/journal.pmed.1001547. Epub 2013 Nov 5. PMID 24223526
- [Result] GBD 2015 Disease and Injury Incidence and Prevalence Collaborators. Global, regional, and national incidence, prevalence, and years lived with disability for 310 diseases and injuries, 1990-2015: a systematic analysis for the Global Burden of Disease Study 2015. Lancet. 2016 Oct 8;388(10053):1545-1602. doi: 10.1016/S0140-6736(16)31678-6. PMID 27733282
- [Result] Machado MO, Veronese N, Sanches M, Stubbs B, Koyanagi A, Thompson T, Tzoulaki I, Solmi M, Vancampfort D, Schuch FB, Maes M, Fava GA, Ioannidis JPA, Carvalho AF. The association of depression and all-cause and cause-specific mortality: an umbrella review of systematic reviews and meta-analyses. BMC Med. 2018 Jul 20;16(1):112. doi: 10.1186/s12916-018-1101-z. PMID 30025524
- [Result] Evans-Lacko S, Knapp M. Global patterns of workplace productivity for people with depression: absenteeism and presenteeism costs across eight diverse countries. Soc Psychiatry Psychiatr Epidemiol. 2016 Nov;51(11):1525-1537. doi: 10.1007/s00127-016-1278-4. Epub 2016 Sep 26. PMID 27667656
- [Result] Mrazek DA, Hornberger JC, Altar CA, Degtiar I. A review of the clinical, economic, and societal burden of treatment-resistant depression: 1996-2013. Psychiatr Serv. 2014 Aug 1;65(8):977-87. doi: 10.1176/appi.ps.201300059. PMID 24789696
- [Result] Lepine BA, Moreno RA, Campos RN, Couttolenc BF. Treatment-resistant depression increases health costs and resource utilization. Braz J Psychiatry. 2012 Dec;34(4):379-88. doi: 10.1016/j.rbp.2012.05.009. PMID 23429808
- [Result] Sanacora G, Zarate CA, Krystal JH, Manji HK. Targeting the glutamatergic system to develop novel, improved therapeutics for mood disorders. Nat Rev Drug Discov. 2008 May;7(5):426-37. doi: 10.1038/nrd2462. PMID 18425072
- [Result] Sanacora G, Treccani G, Popoli M. Towards a glutamate hypothesis of depression: an emerging frontier of neuropsychopharmacology for mood disorders. Neuropharmacology. 2012 Jan;62(1):63-77. doi: 10.1016/j.neuropharm.2011.07.036. Epub 2011 Aug 3. PMID 21827775
- [Result] Hillhouse TM, Porter JH. A brief history of the development of antidepressant drugs: from monoamines to glutamate. Exp Clin Psychopharmacol. 2015 Feb;23(1):1-21. doi: 10.1037/a0038550. PMID 25643025
- [Result] Newport DJ, Carpenter LL, McDonald WM, Potash JB, Tohen M, Nemeroff CB; APA Council of Research Task Force on Novel Biomarkers and Treatments. Ketamine and Other NMDA Antagonists: Early Clinical Trials and Possible Mechanisms in Depression. Am J Psychiatry. 2015 Oct;172(10):950-66. doi: 10.1176/appi.ajp.2015.15040465. PMID 26423481
- [Result] Hare BD, Ghosal S, Duman RS. Rapid Acting Antidepressants in Chronic Stress Models: Molecular and Cellular Mechanisms. Chronic Stress (Thousand Oaks). 2017 Feb;1:2470547017697317. doi: 10.1177/2470547017697317. Epub 2017 Apr 10. PMID 28649673
- [Result] Rasmussen KG. Has psychiatry tamed the "ketamine tiger?" Considerations on its use for depression and anxiety. Prog Neuropsychopharmacol Biol Psychiatry. 2016 Jan 4;64:218-24. doi: 10.1016/j.pnpbp.2015.01.002. Epub 2015 Jan 10. PMID 25582770
- [Result] Naughton M, Clarke G, O'Leary OF, Cryan JF, Dinan TG. A review of ketamine in affective disorders: current evidence of clinical efficacy, limitations of use and pre-clinical evidence on proposed mechanisms of action. J Affect Disord. 2014 Mar;156:24-35. doi: 10.1016/j.jad.2013.11.014. Epub 2013 Dec 10. PMID 24388038
- [Result] Dwyer JM, Duman RS. Activation of mammalian target of rapamycin and synaptogenesis: role in the actions of rapid-acting antidepressants. Biol Psychiatry. 2013 Jun 15;73(12):1189-98. doi: 10.1016/j.biopsych.2012.11.011. Epub 2013 Jan 4. PMID 23295207
- [Result] Duman RS, Li N, Liu RJ, Duric V, Aghajanian G. Signaling pathways underlying the rapid antidepressant actions of ketamine. Neuropharmacology. 2012 Jan;62(1):35-41. doi: 10.1016/j.neuropharm.2011.08.044. Epub 2011 Sep 2. PMID 21907221
- [Result] Akinfiresoye L, Tizabi Y. Antidepressant effects of AMPA and ketamine combination: role of hippocampal BDNF, synapsin, and mTOR. Psychopharmacology (Berl). 2013 Nov;230(2):291-8. doi: 10.1007/s00213-013-3153-2. Epub 2013 Jun 4. PMID 23732839
- [Result] Reich DL, Silvay G. Ketamine: an update on the first twenty-five years of clinical experience. Can J Anaesth. 1989 Mar;36(2):186-97. doi: 10.1007/BF03011442. PMID 2650898
- [Result] Haas DA, Harper DG. Ketamine: a review of its pharmacologic properties and use in ambulatory anesthesia. Anesth Prog. 1992;39(3):61-8. PMID 1308374
- [Result] Zarate CA Jr, Brutsche N, Laje G, Luckenbaugh DA, Venkata SL, Ramamoorthy A, Moaddel R, Wainer IW. Relationship of ketamine's plasma metabolites with response, diagnosis, and side effects in major depression. Biol Psychiatry. 2012 Aug 15;72(4):331-8. doi: 10.1016/j.biopsych.2012.03.004. Epub 2012 Apr 18. PMID 22516044
- [Result] Stahl SM. Mechanism of action of ketamine. CNS Spectr. 2013 Aug;18(4):171-4. doi: 10.1017/S109285291300045X. PMID 23866089
- [Result] Green SM, Hummel CB, Wittlake WA, Rothrock SG, Hopkins GA, Garrett W. What is the optimal dose of intramuscular ketamine for pediatric sedation? Acad Emerg Med. 1999 Jan;6(1):21-6. doi: 10.1111/j.1553-2712.1999.tb00089.x. PMID 9928972
- [Result] Bonanno G, Giambelli R, Raiteri L, Tiraboschi E, Zappettini S, Musazzi L, Raiteri M, Racagni G, Popoli M. Chronic antidepressants reduce depolarization-evoked glutamate release and protein interactions favoring formation of SNARE complex in hippocampus. J Neurosci. 2005 Mar 30;25(13):3270-9. doi: 10.1523/JNEUROSCI.5033-04.2005. PMID 15800181
- [Result] Li N, Liu RJ, Dwyer JM, Banasr M, Lee B, Son H, Li XY, Aghajanian G, Duman RS. Glutamate N-methyl-D-aspartate receptor antagonists rapidly reverse behavioral and synaptic deficits caused by chronic stress exposure. Biol Psychiatry. 2011 Apr 15;69(8):754-61. doi: 10.1016/j.biopsych.2010.12.015. Epub 2011 Feb 3. PMID 21292242
- [Result] Vasavada MM, Leaver AM, Espinoza RT, Joshi SH, Njau SN, Woods RP, Narr KL. Structural connectivity and response to ketamine therapy in major depression: A preliminary study. J Affect Disord. 2016 Jan 15;190:836-841. doi: 10.1016/j.jad.2015.11.018. Epub 2015 Nov 18. PMID 26630613
- [Result] Berman RM, Cappiello A, Anand A, Oren DA, Heninger GR, Charney DS, Krystal JH. Antidepressant effects of ketamine in depressed patients. Biol Psychiatry. 2000 Feb 15;47(4):351-4. doi: 10.1016/s0006-3223(99)00230-9. PMID 10686270
- [Result] Murrough JW, Iosifescu DV, Chang LC, Al Jurdi RK, Green CE, Perez AM, Iqbal S, Pillemer S, Foulkes A, Shah A, Charney DS, Mathew SJ. Antidepressant efficacy of ketamine in treatment-resistant major depression: a two-site randomized controlled trial. Am J Psychiatry. 2013 Oct;170(10):1134-42. doi: 10.1176/appi.ajp.2013.13030392. PMID 23982301
- [Result] Niciu MJ, Luckenbaugh DA, Ionescu DF, Guevara S, Machado-Vieira R, Richards EM, Brutsche NE, Nolan NM, Zarate CA Jr. Clinical predictors of ketamine response in treatment-resistant major depression. J Clin Psychiatry. 2014 May;75(5):e417-23. doi: 10.4088/JCP.13m08698. PMID 24922494
- [Result] Lapidus KA, Levitch CF, Perez AM, Brallier JW, Parides MK, Soleimani L, Feder A, Iosifescu DV, Charney DS, Murrough JW. A randomized controlled trial of intranasal ketamine in major depressive disorder. Biol Psychiatry. 2014 Dec 15;76(12):970-6. doi: 10.1016/j.biopsych.2014.03.026. Epub 2014 Apr 3. PMID 24821196
- [Result] Shiroma PR, Johns B, Kuskowski M, Wels J, Thuras P, Albott CS, Lim KO. Augmentation of response and remission to serial intravenous subanesthetic ketamine in treatment resistant depression. J Affect Disord. 2014 Feb;155:123-9. doi: 10.1016/j.jad.2013.10.036. Epub 2013 Oct 29. PMID 24268616
- [Result] Murrough JW, Perez AM, Pillemer S, Stern J, Parides MK, aan het Rot M, Collins KA, Mathew SJ, Charney DS, Iosifescu DV. Rapid and longer-term antidepressant effects of repeated ketamine infusions in treatment-resistant major depression. Biol Psychiatry. 2013 Aug 15;74(4):250-6. doi: 10.1016/j.biopsych.2012.06.022. Epub 2012 Jul 27. PMID 22840761
- [Result] Singh JB, Fedgchin M, Daly EJ, De Boer P, Cooper K, Lim P, Pinter C, Murrough JW, Sanacora G, Shelton RC, Kurian B, Winokur A, Fava M, Manji H, Drevets WC, Van Nueten L. A Double-Blind, Randomized, Placebo-Controlled, Dose-Frequency Study of Intravenous Ketamine in Patients With Treatment-Resistant Depression. Am J Psychiatry. 2016 Aug 1;173(8):816-26. doi: 10.1176/appi.ajp.2016.16010037. Epub 2016 Apr 8. PMID 27056608
- [Result] Daly EJ, Singh JB, Fedgchin M, Cooper K, Lim P, Shelton RC, Thase ME, Winokur A, Van Nueten L, Manji H, Drevets WC. Efficacy and Safety of Intranasal Esketamine Adjunctive to Oral Antidepressant Therapy in Treatment-Resistant Depression: A Randomized Clinical Trial. JAMA Psychiatry. 2018 Feb 1;75(2):139-148. doi: 10.1001/jamapsychiatry.2017.3739. PMID 29282469
- [Result] Caddy C, Giaroli G, White TP, Shergill SS, Tracy DK. Ketamine as the prototype glutamatergic antidepressant: pharmacodynamic actions, and a systematic review and meta-analysis of efficacy. Ther Adv Psychopharmacol. 2014 Apr;4(2):75-99. doi: 10.1177/2045125313507739. PMID 24688759
- [Result] McGirr A, Berlim MT, Bond DJ, Fleck MP, Yatham LN, Lam RW. A systematic review and meta-analysis of randomized, double-blind, placebo-controlled trials of ketamine in the rapid treatment of major depressive episodes. Psychol Med. 2015 Mar;45(4):693-704. doi: 10.1017/S0033291714001603. Epub 2014 Jul 10. PMID 25010396
- [Result] Erratum: Acute Antidepressant Effects of Intramuscular Versus Intravenous Ketamine: Erratum. Indian J Psychol Med. 2015 Jul-Sep;37(3):379. doi: 10.4103/0253-7176.162911. PMID 26664100
- [Result] aan het Rot M, Collins KA, Murrough JW, Perez AM, Reich DL, Charney DS, Mathew SJ. Safety and efficacy of repeated-dose intravenous ketamine for treatment-resistant depression. Biol Psychiatry. 2010 Jan 15;67(2):139-45. doi: 10.1016/j.biopsych.2009.08.038. PMID 19897179
- [Result] Loo CK, Galvez V, O'Keefe E, Mitchell PB, Hadzi-Pavlovic D, Leyden J, Harper S, Somogyi AA, Lai R, Weickert CS, Glue P. Placebo-controlled pilot trial testing dose titration and intravenous, intramuscular and subcutaneous routes for ketamine in depression. Acta Psychiatr Scand. 2016 Jul;134(1):48-56. doi: 10.1111/acps.12572. Epub 2016 Mar 30. PMID 27028832
- [Derived] Cigognini MA, Guirado AG, van de Meene D, Schneider MA, Salomon MS, de Alexandria VS, Adriano JP, Thaler AM, Fernandes FDS, Carneiro A, Moreno RA. Intramuscular ketamine vs. escitalopram and aripiprazole in acute and maintenance treatment of patients with treatment-resistant depression: A randomized double-blind clinical trial. Front Psychiatry. 2022 Jul 22;13:830301. doi: 10.3389/fpsyt.2022.830301. eCollection 2022. PMID 35935445